CLINICAL TRIAL: NCT05631808
Title: Effect of Epicardial Adipose Tissue Volume and Attenuation on Clinical Outcomes After Acute Ischemic Stroke
Brief Title: Epicardial Adipose Tissue Volume and Attenuation in Acute Ischemic Stroke
Acronym: EATVAS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Other Study IDs: XJTU1AF2022LSK-348
Record Dates: First submitted 2022-11-21; First posted 2022-11-30 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-04

CONDITIONS: Ischemic Stroke
Keywords: Ischemic stroke; Epicardial adipose tissue; Obesity
MeSH Terms: conditions — Ischemic Stroke; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Lowest tertile: Participants with lowest tertile of EAT volume or attenuation among all eligible participants.
  Interventions: Other: Epicardial adipose tissue volume and attenuation
- Intermediate tertile: Participants with intermediate tertile of EAT volume or attenuation among all eligible participants.
  Interventions: Other: Epicardial adipose tissue volume and attenuation
- Highest tertile: Participants with highest tertile of EAT volume or attenuation among all eligible participants.
  Interventions: Other: Epicardial adipose tissue volume and attenuation

INTERVENTIONS:
Other: Epicardial adipose tissue volume and attenuation — Epicardial adipose tissue volume and attenuation assessed by CT are the exposure factors in this study.

SUMMARY:
Excessive accumulation or abnormal distribution of adipose tissue is a recognized risk factor for ischemic stroke. However, the impact of overweight or obesity on clinical outcomes of ischemic stroke is uncertain. The proposition of obesity paradox in stroke patients makes secondary prevention ambiguous for patients with ischemic stroke and overweight or obesity. Body mass index (BMI) or abdominal visceral fat area was used to measure obesity in previous studies. Epicardial adipose tissue (EAT) is a unique visceral fat, which has higher expression of proinflammatory genes than subcutaneous fat and abdominal visceral fat. And inflammation is closely related to the prognosis of ischemic stroke. In this study, the investigators assume EAT volume or attenuation evaluated by chest computed tomography (CT) scan might affect the prognosis of patients with acute ischemic stroke (AIS). Patients with the first acute ischemic stroke will be stratified into tertile groups based on EAT volume or attenuation. The primary endpoint measure is the proportion of patients with a favorable recovery of nerve function deficiency assessed by Modified Rankin Scale （mRS≤2） at 90 days after the onset of symptoms. Secondary endpoints include the following: the percentage of functional recovery measured by the Barthel Index (BI) at day 90 after stroke onset, the propotion of clinical improvement (with an improvement of ≥ 4 points on the National Institute of Health Stroke Scale score or the resolution of the neurologic deficit) or neurological deterioration (with a decline by ≥ 4 points in the total National Institute of Health Stroke Scale score) at day 7 after stroke onset, incidence of hemorrhagic transformation and mortality within 7 days of symptom onset.

ELIGIBILITY:
Inclusion Criteria:

* Patient is between 18 and 80 years of old;
* Acute ischemic stroke（AIS）is diagnosed by brain imaging, and this is the first ischemic stroke event;
* Patient is admitted to hospital within 72 hours after stroke onset;
* Modified Rankin scale score (mRS) ≤2 before onset;
* Patient undergoes chest CT scanning during hospitalization;
* Provision of written informed consent.

Exclusion Criteria:

* Pregnant or nursing women;
* Complicated with cerebral hemorrhage showed by cranial CT on admission;
* Patient had brain tumor, intracranial aneurysm, arteriovenous malformation, or cerebral hemorrhage or underwent brain surgery in the past;
* Severe cardiac, liver, pulmonary, or kidney disease, malignancy, severe coagulation dysfunction, and systemic organ dysfunction;
* Failure to accomplish 7-day and 3-month follow up.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study intends to recruit 200 patients with the first acute ischemic stroke. They undergo chest CT scanning during hospitalization to evaluate epicardial adipose tissue volume and attenuation.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-02-06 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Modified Rankin scale (mRS) | 90 days after stroke onset.
  Assess patients' prognosis by the score of modified Rankin Scale. In the mRS, the lowest score is 0, the highest score is 6, and higher scores mean worse outcome. A score of 0 indicates the patients have no symptoms at all, and a score of 6 indicates the patients are dead. In this study, we evaluate patient's outcomes by the following criteria. A favorable outcome is defined as an mRS score of 0 to 2, an excellent outcome is defined as an mRS score of 0 to 1, whereas a poor outcome is defined as mRS>2.

SECONDARY OUTCOMES:
Barthel Index (BI) | 90 days after stroke onset.
  The percentage of functional recovery from baseline to 90 days after stroke onset, is measured by the Barthel Index (BI). BI score from 0-100, higher scores mean better outcome. We measure how many patients achieve 95 for the BI.
The change of NIHSS score | 7 days after stroke onset.
  The percentage of functional recovery or deterioration from baseline to 7 days after stroke onset, is measured by the National Institute of Health Stroke Scale, short for NIHSS. NIHSS score from 0-42, higher scores mean worse outcome. We define early functional improvement as an improvement of ≥ 4 points on the NIHSS or the resolution of the neurologic deficit, and early neurological deterioration as a decline by ≥ 4 points in the total NIHSS score within 7 days of symptom onset.
Hemorrhagic transformation | within 7 days of symptom onset
  Hemorrhagic transformation is considered present when follow-up MRI or CT scans reveal findings consistent with a newly developed extravasation of blood. Symptomatic intracranial hemorrhage is defined as extravascular blood in the brain confirmed by neuroimaging and is associated with neurological deterioration of ≥ 4 points on the NIHSS.
Mortality | within 7 days of symptom onset
  We evaluate early mortality due to any cause within 7 days of symptom onset.

CONTACTS AND LOCATIONS:
Overall Officials: Guogang Luo, MD, PhD, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Yes